CLINICAL TRIAL: NCT04852146
Title: Electronic Feedback for the Restitution and Valorization of Data on the Management of Acute Coronary Syndrome With ST Segment Elevation in Aquitaine to Emergency Teams
Brief Title: Electronic Feedback for Data Restitution and Valorization to the Emergency Teams in Aquitaine.
Acronym: FERVEUR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Reanim (Unknown); Acira (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/64
Record Dates: First submitted 2021-04-15; First posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Acute Coronary Syndrome
Keywords: electronic feedback; ST+ ACR; Cardiovascular registry
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Professional: The sample of professionals will be made up of doctors and nurses of the emergency structures (pre and intra-hospital), doctors and nurses of interventional cardiology and ambulance drivers practising in an establishment of the 7 participating SAMU zones
  Interventions: Procedure: Electronic feedback
- Patient: The patient sample will consist of patients included in the REANIM registry during the study period (the entire period of the stepped wedge randomised controlled trial).
  Interventions: Procedure: Electronic feedback

INTERVENTIONS:
Procedure: Electronic feedback — Feedbacks have been identified as one of the most effective interventions to improve practices and organisations in health care institutions. It is also a tool for facilitating and coordinating practice registers, improving the contribution of data producers and the quality of data.

SUMMARY:
ST+ Acute Coronary Syndrome (ACS) is a major cause of mortality, morbidity and healthcare costs in Europe and France. Emergency trans-luminal angioplasty (TLA), the gold standard treatment, is the major determinant of vital prognosis and functional recovery of patients with ST+ ACS.

However, data from surveys and French practice registers highlight frequent deviations from the recommendations at different stages of the procedure; in the pre-hospital phase these malfunctions result in longer delays. Improving the quality of care for patients with ST+ ACS, and in particular improving compliance with recommended delays in the acute phase, is a public health priority in France.

Feedback has been identified as one of the most effective interventions to improve practices and organisations in healthcare institutions. Feedbacks are defined as "any summary of a care performance over a given period of time that can be transmitted a posteriori to the health professional in any form, whether written, oral or by computer (in this case called e-feedbacks)". Feedbacks, by objectifying the level of individual and collective performance, encourage recipients to modify their practices and organisations to improve their performance. It also acts as a social pressure mechanism. While the minimum elements of feedback have been identified in the literature, there is a lack of information about the optimal operational modalities for their deployment, which limits the system's capacity to implement them. To overcome this lack of information, there is a consensus in the scientific community that research on feedback should focus not only on analysing its effectiveness, but above all on the determinants of its effectiveness. With regard to the quality of management of patients with ST+ ACS, only four trials were found in the literature that studied the effectiveness of feedbacks; none of them defined the optimal intervention for deploying feedbacks in the emergency department setting.

Practice registers, particularly in the cardiovascular field, have shown their effectiveness in improving practices, particularly through the implementation of feedback to practitioners, who produce data. In 2012, the ARS Aquitaine set up two regional cardiovascular registers constituting permanent, nominative, continuous and exhaustive records of the management of patients suffering from coronary pathologies: the Aquitaine Interventional Cardiology Register (ACIRA) and the Aquitaine Register of Initial Management of Myocardial Infarction (REANIM). The cross-referencing of the REANIM and ACIRA registers constitutes an exhaustive cohort of patients with ST+ ACS containing information on the management of the entire care pathway, from the onset of symptoms to the end of the hospitalization for the management of the acute episode. This cohort, which is unique in France in the field of coronary pathologies, makes it possible to produce unprecedented and highly accurate information, particularly concerning the time taken to provide care. Wishing to actively engage in a process of changing practices, the Aquitaine Cardiovascular Registries team has developed an e-feedback tool for emergency, EMS and cardiology teams. This tool alone cannot contribute to effectively improving patient care. It is necessary to build an intervention for the deployment of this tool that takes into account the scientific data and the organisational constraints of care. Secondly, the evaluation of the effectiveness and economic impact of this e-feedbacks tool deployment intervention will allow us to know its real added value on practices, organisations and health care expenditure.

DETAILED DESCRIPTION:
The study has two phases:

* A phase of construction of the intervention based on qualitative analyses of the focus groups near the professionals of the establishments of the 7 zones SAMU concerned and semi-directive interviews near the directions of the establishments of the 7 zones SAMU concerned;
* A phase of evaluation of the impact of the intervention which is based on a mixed method mixing quantitative and qualitative analyses. The qualitative analyses are based on semi-directive interviews with the professionals concerned in the establishments of the 7 participating UAS zones. The study design of the quantitative part is a cluster randomised controlled trial in a transverse stepped wedge design. The clusters are represented by 7 UAS zones of the ex-Aquitaine region.

ELIGIBILITY:
Patient criteria:

Inclusion Criteria:

* Patients over 18 years of age residing in metropolitan France;
* Patients with ST+ ACS less than 24 hours old;
* Patients treated by one of the 19 SMURs (primary and secondary) or one of the 32 emergency services in Aquitaine.

Exclusion Criteria:

- refusal to participate to REANIM or ACIRA registers.

Professional criteria:

Inclusion Criteria:

- Professionals who volunteered to participate in the interviews, from establishments in the 7 participating emergency zones taking care of patients with ST+ ACS in Ex-Aquitaine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with ST+ ACS, who accept to participate to REANIM or ACIRA registers, and treated by one of the 7 participating emergency zones.
  Professional who volunteered to participate in the interviews,from establishments in the 7 participating emergency zones taking care of patients with ST+ ACS in Ex-Aquitaine.
Sampling Method: Non-Probability Sample
Enrollment: 820 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Assessing effectiveness of an e-feedback deployment intervention. | 28 months after the baseline
  To assess the effectiveness of an e-feedbacks deployment intervention on the proportion of patients with ST+ ACS managed within the recommended time from qualifying ECG to balloon inflation.

SECONDARY OUTCOMES:
Studying acceptability and effectiveness determinants of an e-feedback deployment intervention. | 28 months after the baseline
  Qualitative analysis of acceptability and effectiveness determinants of an e-feedback deployment intervention in emergency facilities: understanding the implementation contexts, usual professionals behaviours, difficulties encountered in practice, needs and expectations with regard to the intervention. Thanks to indicivuals interviews.
Evaluate effectiveness of e-feedback deployment intervention | 28 months after the baseline
  Evaluate effectiveness of e-feedback deployment intervention, thanks to the time between qualifying ECG and balloon inflation
Economic assessment | 28 months after the baseline
  Total cost (in €) of production (design, implementation) of the electronic feedback intervention, thanks to micro-costing
Assessment of health care consumption | 28 months after the baseline
  Difference in health care consumption between the period with and without the intervention and typology of health care consumption between the groups based on SNDS data.

CONTACTS AND LOCATIONS:
Overall Officials: Florence SAILLOUR-GLENISSON, Dr, Study Chair — UMES
Locations (7):
- France (7):
  - Centre Hospitalier Agen Nérac, Agen
  - Centre Hospitalier de la Cote Basque, Bayonne
  - Hôpital Pellegrin, Bordeaux
  - Hôpital de Libourne, Libourne
  - Centre Hospitalier de Mont de Marsan, Mont-de-Marsan
  - Centre Hospitalier de Pau, Pau
  - Centre Hospitalier Périgueux, Périgueux